CLINICAL TRIAL: NCT07180797
Title: Proficiency-Based Progression on Hugo Ras Robot for Learning Nerve-Sparing RARP: Feasibility Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Orsi Academy (Other)
Responsible Party: Sponsor
Other Study IDs: PBP feasibility - RARP - Hugo
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Training Effectiveness
Keywords: surgery; training; robotic assisted surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Robotic-naive participants: urology residents
- Group 2: Intermediate participants: Urologists or urology residents with generic robotic experience using the Intuitive platform, but no exposure to the Hugo system
- Group 3: Experienced participants: Experienced robotic consultants in RARP using the Intuitive platform, but no prior experience with the Hugo system.

SUMMARY:
Feasibility study

1. To evaluate the feasibility of PBP training for nerve-sparing RARP on the Hugo Ras system
2. To assess time to proficiency for participants with varying experience
3. To identify challenges in PBP RARP training through observed errors and feedback

DETAILED DESCRIPTION:
As robotic surgery advances, the emergence of new platforms such as the Hugo™ Robotic-Assisted Surgery System calls for robust training frameworks. Proficiency-Based Progression (PBP) provides a structured method to ensure skill acquisition through clearly defined, measurable benchmarks. This study evaluates the feasibility of implementing a PBP curriculum to train urologists in nerve-sparing robot-assisted radical prostatectomy (RARP) using the Hugo™ system.

Twelve urologists and urology residents will participate, divided into three groups based on experience:

Robotic-naïve Intermediate (Da Vinci experience only) Expert RARP surgeons (Da Vinci experience without prior Hugo exposure)

The PBP training pathway comprises:

Cognitive modules (e-learning with MCQ validation) Psychomotor skills training (device familiarization and basic surgical skills) Procedural training (nerve-sparing RARP on porcine models)

Performance will be evaluated both in real time and via blinded video review.

Primary endpoints include the time to reach proficiency in basic skills and procedural steps, analyzed by prior experience. Secondary endpoints encompass error profiles, participant and instructor feedback, and the feasibility of standardizing proficiency metrics.

ELIGIBILITY:
Inclusion Criteria:

* We'll only include urologist or urology residents to ensure that they have all the same interest and area of expertise

Exclusion Criteria:

Prior experience with the Hugo robotic system. Participants unable to attend all training days. Non-urology residents or consultants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: urology residents and urologists
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
time-to-proficiency for basic skills and procedural steps | 9 months
  * Time taken to achieve proficiency in basic robotic skills on the Hugo system.
  * Time taken to achieve proficiency in RARP using the Hugo system in the simulated setting.

SECONDARY OUTCOMES:
Error patterns and feasibility of PBP RARP training on the Hugo system | 9 months
  Identification of challenging steps/phases in the PBP RARP procedure based on:
  Number of errors committed Feedback from trainers Participant feedback on the training process (structured questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, Professor, Principal Investigator — Orsi Academy
Locations (1):
- Orsi Academy, Melle, Belgium

IPD SHARING:
Plan to Share IPD: No